CLINICAL TRIAL: NCT03110796
Title: Assessment of the Efficacy and Safety of a New Medical Device in the Local Treatment of Diabetic Foot Ulcers: a Prospective, Randomized, Controlled, Double-blind, European Multicentre Clinical Trial
Brief Title: Assessment of the Efficacy and Safety of a New Medical Device in the Local Treatment of Diabetic Foot Ulcers
Acronym: DISCOVERY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FI-16-03-310 3209
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Bandages

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LU3103209 Dose 1 (Experimental): Dressing with LU3103209 Dose 1
  Interventions: Device: Dressing with LU3103209 - Dose 1
- LU3103209 Dose 2 (Experimental): Dressing with LU3103209 Dose 2
  Interventions: Device: Dressing with LU3103209 - Dose 2
- No LU3103209 (Placebo Comparator): Dressing without LU3103209
  Interventions: Device: Dressing without LU3103209

INTERVENTIONS:
Device: Dressing with LU3103209 - Dose 1 — Dressing with LU3103209 - Dose 1
  Arms: LU3103209 Dose 1
Device: Dressing with LU3103209 - Dose 2 — Dressing with LU3103209 - Dose 2
  Arms: LU3103209 Dose 2
Device: Dressing without LU3103209 — Dressing without LU3103209
  Arms: No LU3103209

SUMMARY:
Evaluation of the efficacy and safety of a device with LU3103209 compound versus the same device, free of LU3103209 compound, in the local management of DFUs.

DETAILED DESCRIPTION:
A European prospective, randomized, double-blind, multicentre, clinical trial, conducted in three parallel groups, to evaluate the efficacy and safety of a device with LU3103209 compound versus the same device, free of LU3103209 compound, in the local management of diabetic foot ulcers (DFUs).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years old who has provided his/her written informed consent
2. Patient with Type 1 or Type 2 diabetes mellitus with glycated haemoglobin (HbA1c) level ≤ 10%
3. Inpatient or outpatient who can be monitored by the same investigating team throughout the entire study
4. Patient who agrees to wear an off-loading system during the trial
5. Diagnosis of peripheral neuropathy
6. Patient with an adequate arterial perfusion of the affected limb, confirmed by ABPI and Toe Blood Pressure assessment
7. DFU Grade 1-A or 2-A or 1-C or 2-C as defined by the University of Texas Diabetic Wound Classification System
8. Target DFU surface area between 1 cm² to 10 cm², after debridement
9. DFU present since less than 24 months

Exclusion Criteria:

A. Pregnant or breast-feeding woman or woman of childbearing potential not protected by an effective contraceptive method of birth control B. Patient who participated in another clinical trial in the previous month or who will take part in another clinical trial during the 12 weeks following the inclusion C. Patient with severe renal impairment D. Patient who has presented, during the 3 months before inclusion, an acute ischemic event (acute myocardial infarction or stroke) E. Patient with an active neoplastic condition, treated by radiotherapy, chemotherapy, hormone therapy or immunosuppressant F. Patient treated for a chronic disease requiring high doses of systemic corticosteroids on a daily basis (≥ 40 mg prednisolone) G. Patient with infection which is not controlled by a suitable antibiotic treatment H. Patient with any known allergy or reported adverse reaction to the trial device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
% of Wound Area Regression (WAR), as a measure of efficacy | 12 weeks
  Efficacy of dressings with LU3103209 versus dressing without LU3103209

CONTACTS AND LOCATIONS:
Locations (6):
- Pr JIRKOVSKA, Prague, Czechia
- Pr PETIT, Dijon, France
- Pr PIAGGESI, Pisa, Italy
- Dr KORZON, Gdansk, Poland
- Pr LAZARO, Madrid, Spain
- Pr EDMONDS, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No